CLINICAL TRIAL: NCT06490809
Title: Examining the Clinical Significance of the Change in Manual Dexterity of Parkinson's Patients Receiving Conventional Physiotherapy
Brief Title: Minimal Clinically Important Difference of the Box and Block Test in Parkinson
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emre Şenocak (Other)
Responsible Party: Sponsor-Investigator, Emre Şenocak, Research Assisstant, Karadeniz Technical University
Organization: Karadeniz Technical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: E-13562490-050.01.04-51
Record Dates: First submitted 2024-06-26; First posted 2024-07-08 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Parkinson Disease
Keywords: Parkinson; Box and Block Test; Minimal Clinically Important Difference
MeSH Terms: conditions — Parkinson Disease | interventions — Physical Therapy Modalities

STUDY DESIGN:
Masking Description: An independent Researcher will perform a statistical analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Routine Physiotherapy Group (Experimental): No action will be taken by the researchers on this group's treatment program.
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Physiotherapy — Parkinson's upper extremity rehabilitation generally consists of stretching, strengthening, coordination, recreational activities and skill activities. Exercises will be prescribed by the clinical specialist physician and physiotherapist.

SUMMARY:
The aim of this study is to examine the level of clinical change in gross manual skills of Parkinson's patients who receive conventional physiotherapy. For this purpose, the Box-Block Test will be used, and the amount of change that must occur in the patient's hand functions will be determined for the test to be considered clinically meaningful.

Patients will continue their routine physical therapy sessions and the researchers will not interfere with this program. The treatment program will be created by the clinical specialist physician and physiotherapist.

Upper extremity rehabilitation programs for Parkinson's patients generally consist of methods such as stretching, strengthening, reaching, coordination and recreational activities. Patients will receive physiotherapy for 30 sessions.

ELIGIBILITY:
Inclusion Criteria:

* Being Hoehn & Yahr Stage between 1-3,
* Individuals in the "On" phase,
* Those who were not exposed to any physiotherapy intervention during the initial assessment

Exclusion Criteria:

* Mini-mental status assessment < 24 points;
* Presence of severe dyskinesia,
* Those who experience fluctuations in the on-off phase,
* Those who have undergone stereotaxic brain surgery for Parkinson's,
* Individuals with changes in dopamine dose within three months,
* Presence of unstable cardiac and respiratory disease
* Those with an orthopedic problem or a history of surgery affecting upper extremity performance.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Box and Block Test | Baseline of the study
  This test assesses gross manual dexterity. The number of wooden blocks moved during 60 seconds gives the total score. A high score indicates good dexterity.
Box and Block Test | 6 weeks (5 session days for 6 weeks)
  This test assesses gross manual dexterity. The number of wooden blocks moved during 60 seconds gives the total score. A high score indicates good dexterity.
Global Rating of Patient-Perceived Changes (GRP-PC) | 6 weeks (5 session days for 6 weeks)
  GRP-PC will used to assess patient-perceived hand dexterity changes after the routine intervention. The patient will first asked, "Has your hand dexterity changed compared to when you did not receive interventions?". If the answer is no, the person will given a score of 0 (i.e. no change). In the case of positive response, the patient will asked, "How much better or worse is your hand dexterity" and the patient response will scored on the following 14-point Likert scale: +7 (very much better), +6 (much better), +5 (better), +4 (relatively better), +3 (somewhat better), +2 (a little better), +1 (very little better), -1 (very little worse), -2 (a little worse), -3 (somewhat worse), -4 (relatively worse), -5 (worse), -6 (much worse), and -7 (very much worse). This form will only be used to classify patients' satisfaction with treatment at the end of the study.

SECONDARY OUTCOMES:
Demographic Data Form | Baseline of the study
  This form was created by researchers and it consist of personal informations such as gender, education, age, body mass index, dominant and affected extremity, disease duration, using medicine

CONTACTS AND LOCATIONS:
Overall Officials: Murat Emirzeoğlu, PhD, Study Chair — Karadeniz Technical University; Tuğba Eyigürbüz, PhD, Study Chair — Bağcılar Education and Research Hospital; Adem Aktürk, PhD, Study Chair — İstanbul Gelişim University
Locations (1):
- Özel Öz İstanbul Tıp Merkezi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided